CLINICAL TRIAL: NCT00378326
Title: Immunotherapy of the Paraneoplastic Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDA-0572
Record Dates: First submitted 2006-09-18; First posted 2006-09-20 (Estimated); Results first posted 2016-02-23 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Paraneoplastic Syndromes
Keywords: paraneoplastic syndrome
MeSH Terms: conditions — Paraneoplastic Syndromes | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus (Experimental): Tacrolimus at doses of 0.15- 0.3mg/kg/day in two divided oral doses, in conjunction with, initially, up to 60mg/day of oral prednisone
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus at doses of 0.15- 0.3mg/kg/day in two divided oral doses, in conjunction with, initially, up to 60mg/day of oral prednisone
  Other Names: FK506

SUMMARY:
We treat a subset of patients with paraneoplastic neurologic disorders, including those with Yo-mediated paraneoplastic cerebellar degeneration (PCD), the Hu syndrome, which is most commonly associated with small cell lung cancer (SCLC) - paraneoplastic subacute sensory neuropathy, encephalomyelitis, limbic encephalopathy, autonomic neuropathy - and the Ri Syndrome (a.k.a. Paraneoplastic Opsoclonus-Myoclonus Ataxia), as well as those patients suspected to have a paraneoplastic neurologic disorder but in whom a characteristic antibody has not yet been identified. Our treatment protocol consists of immune suppression therapy using tacrolimus (FK506), a potent inhibitor of lymphocyte proliferation that is commonly used to prevent organ transplant rejection.

DETAILED DESCRIPTION:
Patients may stay either in-hospital while being treated with Tacrolimus, receive treatment as an outpatient, or a combination of the two. Additionally, patients who are too sick to be treated at Rockefeller University (RU) (eg. patients actively seizing), but are in need of urgent treatment, may be treated at either Memorial Sloan-Kettering Cancer Center or New York-Presbyterian Hospital. During treatment, patients will undergo blood draws, at set intervals (see section g below), clinical evaluation, possibly repeat leukapheresis or large volume blood draw, and lumbar puncture (see below). Since many patients live far away from New York, some of these procedures may be performed by RU staff or in conjunction with their local MDs.

Patients who are terminated from Tacrolimus treatment after 7-21 days will be followed up as outpatients for evaluation of their neurologic and medical status. Wherever possible, these patients will be seen on days 3 and 10 post treatment termination, and then on a biweekly basis for two months. Since many patients live far away from New York, they may instead be monitored in conjunction with their local MDs. Patients who show a definite clinical response to Tacrolimus may be maintained on a therapeutic dose for up to one year, and will be followed as outpatients. For patients receiving retreatment, they may be treated as inpatients or on an outpatient basis, at the discretion of the PI, on the same schedule as patients being treated initially. Long term improvement or decline in neurologic function will be objectively assessed by neurologic exam, which will be quantified by use of the Karnofsky scale (a measure of functional neurologic status). Since the vast majority of Hu patients decline over a 6-12 month period following diagnosis, a stable or improved Karnofsky score over such a time period will be taken as a measure of successful treatment. Repeat lumbar puncture (up to eight per year) and leukapheresis or large volume blood draw (approx. 100 cc) may be performed (up to four of each per year), especially in the setting of neurologic change, to assess the immune responses to the medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Paraneoplastic Disorder

Exclusion Criteria:

* Metastasis (spread) of cancer to brain, History of additional active malignancy other than non-melanoma skin cancer, History of Hepatitis B, Hepatitis C, HIV or Syphilis.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Darnell, MD, PhD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- [Derived] Orange D, Frank M, Tian S, Dousmanis A, Marmur R, Buckley N, Parveen S, Graber JJ, Blachere N, Darnell RB. Cellular immune suppression in paraneoplastic neurologic syndromes targeting intracellular antigens. Arch Neurol. 2012 Sep;69(9):1132-40. doi: 10.1001/archneurol.2012.595. PMID 22566506

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tacrolimus
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tacrolimus
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 59.5 [31 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 1

OUTCOME MEASURES:

1. Secondary Outcome: Cerebrospinal Fluid (CSF) Pleocytosis
Time Frame: White blood cell count in CSF was measured at two time points, pre- and post-treatment
Population: 19 treatment events in 16 patients at which both pre- and post-treatment CSF samples available.
  The data are reported below, separately for pre-treatment samples and post-treatment samples.
Measure: Median (Full Range); unit: cells/mm^3
Units Other Than Participants: Treatment events
Groups:
- Pre-treatment: White blood cell (WBC) count in CSF pre-treatment
- Post-treatment: White blood cell (WBC) count in CSF post-treatment
Arm/Group | Pre-treatment | Post-treatment
Number analyzed (Participants) | 16 | 16
Number analyzed (Treatment events) | 19 | 19
cells/mm^3 | 3 [0 to 51] | 3 [0 to 41]

2. Primary Outcome: Survival of Patients With Paraneoplastic Disease Who Are Treated With Tacrolimus
Description: Survival in patients with paraneoplastic disease who are treated with Tacrolimus, from time of tacrolimus treatment
Time Frame: through study completion, median 3 years of follow up
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Tacrolimus: Tacrolimus at doses of 0.15-0.3mg/kg/day in two divided oral doses, in conjunction with, initially, up to 60mg/day of oral prednisone
Arm/Group | Tacrolimus
Number analyzed (Participants) | 26
months | 48 [22 to 72]

ADVERSE EVENTS:
Groups:
- All Patients: All patients enrolled
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 3/26
Other Adverse Events (participants affected / at risk) | 10/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=26)
Hospitalization, search for primary tumor (Surgical and medical procedures) | 1 (1)
Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ataxia and weakness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=26)
Albumin, serum low (General disorders) | 3 (3)
ALT, serum high (General disorders) | 1 (1)
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
AST, serum high (General disorders) | 1 (1)
BUN, serum high (General disorders) | 4 (6)
calcium, serum low (General disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)
dizziness (General disorders) | 1 (1)
swallowing difficulty (Gastrointestinal disorders) | 1 (1)
glucose, serum high (General disorders) | 5 (6)
HCT, low (Blood and lymphatic system disorders) | 3 (3)
headache (General disorders) | 3 (3)
hgb, low (Blood and lymphatic system disorders) | 4 (4)
dysarthria (Nervous system disorders) | 1 (1)
tremor (Nervous system disorders) | 3 (5)
insomnia (General disorders) | 1 (1)
hot flashes (General disorders) | 1 (1)
lymphocytes, low (Blood and lymphatic system disorders) | 1 (1)
depression (General disorders) | 1 (1)
neutrophils, high (Blood and lymphatic system disorders) | 1 (1)
numbness/tingling (Nervous system disorders) | 1 (1)
platelets, low (Blood and lymphatic system disorders) | 1 (1)
potassium, serum high (General disorders) | 1 (1)
potassium, serum low (General disorders) | 2 (2)
PTT, high (General disorders) | 2 (2)
RBC low (Blood and lymphatic system disorders) | 4 (4)
blurred vision (General disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
WBC high (Blood and lymphatic system disorders) | 2 (2)
WBC, low (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes